CLINICAL TRIAL: NCT03287609
Title: EVOlocumab for Early Reduction of LDL-cholesterol Levels in Patients With Acute Coronary Syndromes (EVOPACS) - A Randomized, Double-blind, Placebo-controlled Multicenter Study
Brief Title: EVOlocumab for Early Reduction of LDL-cholesterol Levels in Patients With Acute Coronary Syndromes (EVOPACS)
Acronym: EVOPACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Amgen (Industry); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-01753
Record Dates: First submitted 2017-09-07; First posted 2017-09-19 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evolocumab (Active Comparator): Evolocumab 140 mg/mL, pre-filled auto-injector pen, 3 injections at day 1 and week 4
  Interventions: Drug: Evolocumab 140 mg/mL
- Placebo (Placebo Comparator): Placebo, pre-filled auto-injector pen, 3 injections at day 1 and week 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab 140 mg/mL — Three injections with pre-filled auto-injector pen at day 1 and at week 4.
  Arms: Evolocumab
Drug: Placebo — Three injections with pre-filled auto-injector pen at day 1 and at week 4.
  Arms: Placebo

SUMMARY:
Reduction of low-density lipoprotein cholesterol (LDL-C) levels effectively reduces the risk of adverse events in patients with established atherosclerotic cardiovascular disease. The clinical benefit of statins in improving clinical outcomes is proportional to the magnitude of LDL-C reduction, is more pronounced in patients with acute coronary syndromes (ACS) compared with stable coronary artery disease, and emerges at very early stages (as early as 4 weeks) after ACS when statins are administered in the acute phase of the event. On the basis of this evidence, early initiation of statin therapy is currently recommended in patients presenting with ACS. Because many patients cannot achieve adequate reduction of LDL-C levels despite treatment with high doses of statins or non-statin lipid-modifying medications, substantial residual risk remains. Moreover, the time of onset of LDL-C reduction takes 2 weeks following initiation of statin therapy. Proprotein convertase subtilisin/kexin type-9 (PCSK9) inhibitors represent a novel class of lipid-lowering drugs leading to rapid, profound, and consistent reductions in LDL-C levels. While the effectiveness of PCSK9 monoclonal antibodies for LDL-C lowering has been established across patient populations without atherosclerotic cardiovascular disease or with stable ischemic heart disease, reduction and attainment of LDL-C target levels has not been explored in the acute setting of ACS - a clinical setting with highest risk of early event recurrence (within the first month). In this study the investigators want to evaluate the safety and effectiveness of the PCSK9 inhibitor evolocumab as compared with placebo, administered in the acute phase of ACS, for reduction of LDL-C levels within 8 weeks in patients receiving guideline-recommended high-intensity statin treatment (atorvastatin 40mg QD).

ELIGIBILITY:
Inclusion Criteria:

Male or female ≥ 18 years of age;

* Hospitalized for a recent ACS;
* LDL-C levels defined as follows:
* LDL-C ≥70 mg/dL (≥1.8 mmol/L) or non-HDL-C ≥100 mg/dL (≥2.6 mmol/) in patients who have been receiving stable treatment with high-intensity statin within ≥ 4 weeks prior to enrollment (i.e. continuous treatment that has not changed with regard to statin intensity over the past 4 weeks) or, LDL-C ≥90 mg/dL (≥2.3 mmol/L) or non-HDL-C ≥120 mg/dL (≥3.1 mmol/) in patients who have been receiving stable treatment with low- or moderate-intensity statin within ≥ 4 weeks prior to enrollment (i.e. continuous treatment that has not changed with regard to statin intensity over the past 4 weeks), or LDL-C ≥125 mg/dL (≥3.2 mmol/L) or non-HDL-C ≥155 mg/dL (≥4.0 mmol/) in patients who are statin-naïve or have not been on a stable (unchanged) statin regimen for at least 4 weeks prior to enrollment;
* Ability to understand the requirements of the study and to provide informed consent.

Exclusion Criteria:

* Unstable clinical status (hemodynamic or electrical instability;
* Uncontrolled cardiac arrhythmia, defined as recurrent and symptomatic ventricular tachycardia or atrial fibrillation with rapid ventricular response not controlled by medications in the past 3 months prior to screening;
* Severe renal dysfunction, defined by estimated glomerular filtration rate <30 ml/min/1.73m2;
* Active liver disease or hepatic dysfunction, either reported in patient medical record or defined by asparate aminotransferase (AST) or alanine aminotransferase (ALT) levels > 3x the upper limit of normal;
* Reported intolerance to atorvastatin (any dose) OR statin intolerance;
* Known allergy to contrast medium, heparin, aspirin, ticagrelor or prasugrel;
* Known sensitivity to any substances to be administered;
* Patients who previously received evolocumab or other PCSK9 inhibitor;
* Patient who received cholesterol ester transfer protein inhibitors in the past 12 months prior to screening;
* Treatment with systemic steroids or systemic cyclosporine in the past 3 months systemic cyclosporine, systemic steroids (eg. intravenous, intramuscular or per os);
* Known active infection or major hematologic, metabolic, or endocrine dysfunction in the judgment of the Investigator;
* Patients who will not be available for study-required procedures in the judgment of the Investigator;
* Current enrollment in another investigational device or drug study;
* Active malignancy requiring treatment;
* Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Percent change in calculated LDL-C in the intent to treat (ITT) population | Baseline to week 8

SECONDARY OUTCOMES:
Number of patients with adverse events and serious adverse events | Baseline to week 8

OTHER OUTCOMES:
Nominal change in calculated LDL-C | Baseline to week 8
Proportion of patients with LDL-C level <70 mg/dL (<1.8 mmol/L) at week 8 | Baseline to week 8
Change in total cholesterol in the ITT population | Baseline to week 8
Change in HDL-C in the ITT population | Baseline to week 8
Change in lipoprotein-a in the ITT population | Baseline to week 8
Change in triglycerides in the ITT population | Baseline to week 8
Change in non-HDL-C in the ITT population | Baseline to week 8
Change in apolipoprotein B in the ITT population | Baseline to week 8
Change in apolipoprotein A-1 in the ITT population | Baseline to week 8
Percent change in high-sensitivity CRP (hs-CRP) in the ITT population | Baseline to week 8
Proportion of patients with hs-CRP level <2 mg/dL at week 8 in the ITT population | Baseline to week 8
Proportion of patients with LDL-C <70 mg/dL and hs-CRP <2 mg/dL at week 8 in the ITT population | Baseline to week 8
Nominal change in Interleukin (IL)-1b and IL-6 in the ITT population | Baseline to week 8
Change in high-sensitivity Troponin T | Baseline to 72 hours
Area under the curve (AUC) at Multiplate with Adenosinediphosphate (ADP) test | Baseline to 72 hours and to week 8
  Platelet inhibition assessed with Multiplate ADP test at 72 hours and 8 weeks
Area under the curve (AUC) at Multiplate with Thrombin receptor activating peptide (TRAP) test | Baseline to 72 hours and to week 8
  Platelet inhibition assessed with Multiplate TRAP test at 72 hours and 8 weeks
Number of patients with contrast-induced acute kidney injury (CI-AKI) at 72 hours among patients who undergo coronary angiography at baseline | Baseline to 72 hours
Number of patients with adjudicated events (death, cardiovascular death, myocardial infarction, hospitalization for recurrent ACS, hospitalization for heart failure, coronary revascularization, stroke | Baseline to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Prof., MD, Study Chair — Bern University Hospital; Konstantinos Koskinas, MD, Principal Investigator — Bern University Hospital
Locations (7):
- Switzerland (7):
  - Basel University Hospital, Basel, Canton of Basel-City
  - HFR Kantonsspital, Fribourg, Canton of Fribourg
  - Hopitaux Universitaires Geneve, Geneva, Canton of Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - University Hospital, Zurich, Canton of Zurich
  - Cardiocentro Ticino, Lugano, Canton Ticino
  - Bern University Hospital, Bern

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers

REFERENCES:
- [Result] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Result] Lipinski MJ, Benedetto U, Escarcega RO, Biondi-Zoccai G, Lhermusier T, Baker NC, Torguson R, Brewer HB Jr, Waksman R. The impact of proprotein convertase subtilisin-kexin type 9 serine protease inhibitors on lipid levels and outcomes in patients with primary hypercholesterolaemia: a network meta-analysis. Eur Heart J. 2016 Feb 7;37(6):536-45. doi: 10.1093/eurheartj/ehv563. Epub 2015 Nov 17. PMID 26578202
- [Result] Ray KK, Cannon CP, McCabe CH, Cairns R, Tonkin AM, Sacks FM, Jackson G, Braunwald E; PROVE IT-TIMI 22 Investigators. Early and late benefits of high-dose atorvastatin in patients with acute coronary syndromes: results from the PROVE IT-TIMI 22 trial. J Am Coll Cardiol. 2005 Oct 18;46(8):1405-10. doi: 10.1016/j.jacc.2005.03.077. PMID 16226162
- [Result] Schwartz GG, Olsson AG, Ezekowitz MD, Ganz P, Oliver MF, Waters D, Zeiher A, Chaitman BR, Leslie S, Stern T; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) Study Investigators. Effects of atorvastatin on early recurrent ischemic events in acute coronary syndromes: the MIRACL study: a randomized controlled trial. JAMA. 2001 Apr 4;285(13):1711-8. doi: 10.1001/jama.285.13.1711. PMID 11277825
- [Result] Navarese EP, Kolodziejczak M, Kereiakes DJ, Tantry US, O'Connor C, Gurbel PA. Proprotein Convertase Subtilisin/Kexin Type 9 Monoclonal Antibodies for Acute Coronary Syndrome: A Narrative Review. Ann Intern Med. 2016 May 3;164(9):600-7. doi: 10.7326/M15-2994. Epub 2016 Mar 22. PMID 26999484
- [Derived] Koskinas KC, Windecker S, Pedrazzini G, Mueller C, Cook S, Matter CM, Muller O, Haner J, Gencer B, Crljenica C, Amini P, Deckarm O, Iglesias JF, Raber L, Heg D, Mach F. Evolocumab for Early Reduction of LDL Cholesterol Levels in Patients With Acute Coronary Syndromes (EVOPACS). J Am Coll Cardiol. 2019 Nov 19;74(20):2452-2462. doi: 10.1016/j.jacc.2019.08.010. Epub 2019 Aug 31. PMID 31479722